CLINICAL TRIAL: NCT00914732
Title: Comparison of the Safety and Immunogenicity of Lyophilized IMVAMUNE® (1x10^8 TCID50) Versus Liquid Formulation IMVAMUNE® (1x10^8 TCID50) Administered by the Subcutaneous Route and a Lower Dose Liquid Formulation IMVAMUNE® (2x10^7 TCID50) Administered by the Intradermal Route in Healthy Vaccinia-Naïve Individuals
Brief Title: Lyophilized IMVAMUNE® (1x10^8 TCID50) Versus Liquid IMVAMUNE® (1x10^8 TCID50) Administered Subcutaneously and a Lower Dose Liquid IMVAMUNE® (2x10^7 TCID50) Administered Intradermally
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 09-0002; POX-MVA-029
Record Dates: First submitted 2009-06-04; First posted 2009-06-05 (Estimated); Results first posted 2021-01-12 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2011-01

CONDITIONS: Smallpox
Keywords: IMVAMUNE®, smallpox, vaccine
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- Group B, liquid, subcutaneous (Experimental): Group B: 165 subjects will receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) liquid formulation by the subcutaneous route on Day 0 and 28.
  Interventions: Biological: MVA Smallpox Vaccine
- Group C, liquid, intradermal (Experimental): Group C: 165 subjects will receive a 2 dose regimen of IMVAMUNE® (2x10^7 TCID50/0.1mL per dose) liquid formulation by the intradermal route on Day 0 and 28.
  Interventions: Biological: MVA Smallpox Vaccine
- Group A, lyophilized, subcutaneous (Experimental): Group A: 165 subjects will receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) lyophilized formulation by the subcutaneous route on Day 0 and 28.
  Interventions: Biological: MVA Smallpox Vaccine

INTERVENTIONS:
Biological: MVA Smallpox Vaccine — Vaccinia vaccine liquid formulation delivered by subcutaneous (SC) route at 1x10^8 TCID50 per 0.5 mL dose on Days 0 and 28.
  Arms: Group B, liquid, subcutaneous
Biological: MVA Smallpox Vaccine — Vaccinia vaccine liquid formulation delivered at lower dose [2x10^7 tissue culture infectious dose 50 (TCID50) per 0.1 mL dose] by intradermal (ID) route on Days 0 and 28.
  Arms: Group C, liquid, intradermal
Biological: MVA Smallpox Vaccine — Vaccinia vaccine lyophilized formulation delivered by subcutaneous (SC) route at 1x10^8 TCID50 per 0.5 mL dose on Days 0 and 28.
  Arms: Group A, lyophilized, subcutaneous

SUMMARY:
Due to recent concern of biowarfare and bioterrorism, the US government is making efforts to improve its ability to protect citizens against the smallpox virus. This study will evaluate safety of IMVAMUNE®, an investigational smallpox vaccine, and its ability to stimulate the immune system (the body's defense system). Two vaccine preparations have the same name but one is a liquid and one is a powder that has liquid added just before it is given. The vaccine that comes as a liquid will be injected (given as a shot) just under the skin (subcutaneously) or injected between the layers of the skin (intradermally). The powder formulation is only injected just under the skin. Approximately 495 adults, age 18 older born after 1971, which have not had smallpox vaccine before, may participate in the study for about 7 months.

DETAILED DESCRIPTION:
Smallpox was declared officially eradicated by the World Health Assembly in 1980. Despite the fact that the World Health Organization (WHO) officially declared smallpox to be eradicated, a new threat exists due to the potential use of variola virus as an agent for biological warfare and/or bio-terrorism. Following the events of September 11, 2001 the Division of Microbiology and Infectious Diseases/National Institute of Allergy and Infectious Diseases contracted for the advanced development of IMVAMUNE®. Initially, a lyophilized formulation was manufactured, which was reconstituted 'at the bedside' prior to administration in clinical and non-clinical settings. Due in part to the potential requirement for mass vaccinations coupled with the increased manufacturing time and other constrains associated with lyophilization, it was decided to transition to a liquid product formulation. Therefore, after 2005, clinical and non-clinical efforts have focused largely on the liquid formulation, though non-clinical studies with the lyophilized formulation continued. Presently, due to the potential need to be able to stockpile Modified Vaccinia Ankara (MVA) for an extended period of time, there is renewed interest in the lyophilized formulation. The purpose of this study is to compare the safety and immunogenicity of lyophilized IMVAMUNE® [1x10^8 tissue culture infectious dose 50 (TCID50)] versus liquid formulation IMVAMUNE® (1x10^8 TCID50) administered by the subcutaneous (SC) route and a lower dose liquid formulation IMVAMUNE® (2x10^7 TCID50) administered by the intradermal (ID) route in healthy vaccinia-naïve individuals. This study is designed as a randomized, non-placebo controlled, partially-blinded study (liquid versus lyophilized formulation by the SC route Group B versus A). The study staff is unblinded to Group C. The study will contain 3 arms: Group A [Number (N)=165] will receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) lyophilized formulation by the SC route on Day 0 and 28. Group B (N=165) will receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) liquid formulation by the SC route on Day 0 and 28. Group C (N=165) will receive a 2 dose regimen of IMVAMUNE® (2x10^7 TCID50/0.1 mL per dose) liquid formulation by the ID route on Day 0 and 28. Safety will be measured by assessment of solicited local and systemic reactions within 15 days after each vaccination (Day 0-14), unsolicited adverse events for 28 days following the second vaccination (56 days following the initial vaccination for those subjects that fail to receive the second vaccination), and serious adverse events through six months post the final vaccination. Immunogenicity testing will include assessment of vaccinia-specific plaque reduction neutralizing antibody titers (PRNT) and enzyme linked immunosorbent assay (ELISA) mean geometric titers (GMT) based on individual peak titers. For each subject, the peak PRNT or ELISA will be defined as the largest titer among all available measurements post second vaccination.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria that must be met prior to the initial vaccination:

* At least 18 years of age and born after 1971.
* Read, signed, and dated informed consent document.
* Available for follow-up for the planned duration of the study (6 months after last immunization).
* Acceptable medical history by screening evaluation and limited physical assessment.
* If the subject is female and of childbearing potential, negative serum pregnancy test at screening and negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the subject is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for 28 days following the last vaccination:

  1. A woman is considered of childbearing potential unless post-menopausal (greater than or equal to 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy).
  2. Acceptable contraception methods are restricted to effective devices [intrauterine devices (IUD)s, NuvaRing®] or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus), and monogamous relationship with a vasectomized partner.
* Negative enzyme linked immunosorbent assay (ELISA) for human immunodeficiency virus (HIV).
* Alanine aminotransferase (ALT) <1.25 times institutional upper limit of normal.
* Negative hepatitis B surface antigen and negative antibody to hepatitis C virus.
* Negative urine glucose and urine protein <1 plus by dipstick or urinalysis.
* Adequate renal function is defined as a serum creatinine not exceeding the institution's upper limit of normal.
* Electrocardiogram (ECG) in absence of clinical significance (e.g., complete left or right bundle branch block, incomplete left bundle branch block or sustained ventricular arrhythmia, or 2 premature ventricular contraction's (PVC)'s in a row, or sympathetic tonus (ST) elevation consistent with ischemia).
* The following blood parameters:

  1. Hemoglobin equal or above the lower limit of institutional normal (sex-specific);
  2. White blood cells greater than 2,500 and less than 11,000/mm^3;
  3. Platelets greater than or equal to 140,000/mm^3.
* Weight: greater than or equal to 110 pounds.

Inclusion Criteria that must be met prior to the second vaccination:

* Acceptable medical history.
* If the subject is female and of childbearing potential, negative urine or serum pregnancy test within 24 hours prior to vaccination.
* If the subject is female and of childbearing potential, she agrees to use acceptable contraception, and not become pregnant for 28 days following the last vaccination:

  1. A woman is considered of childbearing potential unless post-menopausal (greater than or equal to 1 year) or surgically sterilized (tubal ligation, bilateral oophorectomy, or hysterectomy).
  2. Acceptable contraception methods are restricted to effective devices (IUDs, NuvaRing®) or licensed hormonal products with use of method for a minimum of 30 days prior to vaccination, abstinence from sexual intercourse with men (vaginal penetration by a penis, coitus), and monogamous relationship with a vasectomized partner.

Exclusion Criteria:

Exclusion criteria that apply prior to the initial vaccination:

* History of immunodeficiency
* Typical vaccinia scar
* Known or suspected history of smallpox vaccination including Modified Vaccinia Ankara (MVA) alone or as a vector as well as other investigational smallpox vaccine
* Military service prior to 1991 or after January 2003
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease, diabetes mellitus, or moderate to severe kidney impairment
* Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site
* Active autoimmune disease

  a. Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor
* Systolic blood pressure greater than or equal to 150 mmHg or diastolic blood pressure greater than or equal to 100 mmHg
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hp2010.nhlbihin.net/atpiii/calculator.asp)

NOTE that this criterion applies only to subjects 20 years of age and older AND only if at least one of the following apply:

a. have smoked a cigarette in the past month, and/or b. have hypertension (defined as systolic blood pressure >140 mm Hg) or are on antihypertensive medication, and/or c. have a family history of coronary heart disease in male first-degree relative (father or brother) <55 years of age or a female first-degree relative (mother or sister) <65 years of age

* High-dose steroid use for greater than 2 weeks duration within three months prior to vaccination and current use of immunosuppressive medication

  1. Corticosteroid nasal sprays are permissible
  2. Persons who are using a topical steroid can be enrolled after their therapy is completed
  3. Inhaled steroids for asthma are not permissible
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* Any history of illegal injection drug use
* Receipt or planned receipt of inactivated vaccine from 14 days prior to the first vaccination through 14 days post second vaccination
* Receipt or planned receipt of any other live attenuated vaccine within 30 days prior to the first vaccination through 30 days post second vaccination
* Use of any other experimental agent within 30 days prior to vaccination and for the duration of the study
* Receipt of blood products or immunoglobulin within six months prior to vaccination
* Donation of a unit of blood within 56 days prior to vaccination and prior to Visit 6
* Acute febrile illness (greater than or equal to 100.4 degrees Fahrenheit) on the day of vaccination
* Pregnant or lactating women
* Eczema of any degree or history of eczema
* Active atopic dermatitis, active exfoliative skin disorders/conditions, current Varicella zoster, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm
* Any condition that, in the opinion of the investigator, might interfere with study objectives
* Known allergy to IMVAMUNE® vaccine
* Known allergy to egg or aminoglycoside (including gentamicin)
* Study personnel

Exclusion criteria that apply prior to the second vaccination:

* Continued inflammation (erythema and/or induration) graded as moderate or severe at the site of the initial vaccination
* History of immunodeficiency
* Known or suspected impairment of immunologic function including, but not limited to, clinically significant liver disease, diabetes mellitus, or moderate to severe kidney impairment
* Malignancy not including squamous cell skin cancer or basal cell skin cancer unless at the vaccination site or history of skin cancer at the vaccination site
* Active autoimmune disease

  a. Persons with vitiligo or thyroid disease (e.g., taking thyroid hormone replacement) are not excluded
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, or other heart condition under the care of a doctor
* Systolic blood pressure greater than or equal to 150 mmHg or diastolic blood pressure greater than or equal to 100 mmHg
* High-dose steroid use for greater than 2 weeks duration within three months prior to vaccination and current use of immunosuppressive medication.

  1. Corticosteroid nasal sprays are permissible
  2. Persons who are using a topical steroid can be enrolled after their therapy is completed
  3. Inhaled steroids for asthma are not permissible
* Medical or psychiatric condition or occupational responsibilities that preclude subject compliance with the protocol
* Any history of illegal injection drug use
* Receipt of or planned receipt of inactivated vaccine from 14 days prior to vaccination through 14 days post second vaccination
* Receipt of or planned receipt of any other live attenuated vaccine from 30 days prior to vaccination through 30 days post second vaccination
* Use of any other experimental agent within 30 days prior to vaccination and for the duration of the study
* Receipt of blood products or immunoglobulin within six months prior to vaccination
* Donation of a unit of blood within 56 days prior to vaccination and prior to Visit 6
* Acute febrile illness (greater than or equal to 100.4 degrees Fahrenheit) on the day of vaccination
* Pregnant or lactating women
* Eczema of any degree or history of eczema
* Active atopic dermatitis, active exfoliative skin disorders/conditions, current Varicella zoster, or any acute skin disorders of large magnitude, e.g., laceration requiring sutures, burn greater than 2×2 cm
* Any condition that, in the opinion of the investigator, might interfere with study objectives
* Known allergy to IMVAMUNE® vaccine
* Known allergy to egg or aminoglycoside (including gentamicin)

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 523 (Actual)
Dates: Start 2010-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Emory Vaccine Center - The Hope Clinic, Decatur, Georgia
  - University of Iowa - Vaccine Research & Education Unit, Iowa City, Iowa
  - University of Maryland School of Medicine - Center for Vaccine Development - Baltimore, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Vanderbilt University Hospital - Pediatric Clinical Research, Nashville, Tennessee
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Group Health Research Institute - Seattle, Seattle, Washington
  - The University of Washington - Virology Research Clinic, Seattle, Washington

REFERENCES:
- [Derived] Frey SE, Stapleton JT, Ballas ZK, Rasmussen WL, Kaufman TM, Blevins TP, Jensen TL, Davies DH, Tary-Lehmann M, Chaplin P, Hill H, Goll JB; DMID 09-0002 MVA Vaccine Study Group. Human Antibody Responses Following Vaccinia Immunization Using Protein Microarrays and Correlation With Cell-Mediated Immunity and Antibody-Dependent Cellular Cytotoxicity Responses. J Infect Dis. 2021 Oct 28;224(8):1372-1382. doi: 10.1093/infdis/jiab111. PMID 33675226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy adults age 18 and older (born after 1971) recruited from existing volunteer populations and from the communities at large around the clinical sites. Participants were enrolled between 09FEB2010 and 02SEP2010.
Groups:
- Lyophilized, Subcutaneous: Participants receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) lyophilized formulation by the subcutaneous route on Day 0 and 28.
- Liquid, Subcutaneous: Participants receive a 2 dose regimen of IMVAMUNE® (1x10^8 TCID50/0.5 mL per dose) liquid formulation by the subcutaneous route on Day 0 and 28.
- Liquid, Intradermal: Participants receive a 2 dose regimen of IMVAMUNE® (2x10^7 TCID50/0.1mL per dose) liquid formulation by the intradermal route on Day 0 and 28.
Period: Overall Study
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous | Liquid, Intradermal
Started | 165 | 167 | 191
Received Second Vaccination | 150 | 157 | 153
Completed | 155 | 160 | 180
Not Completed | 10 | 7 | 11
Not completed — Lost to Follow-up | 6 | 7 | 9
Not completed — Withdrawal by Subject | 3 | 0 | 2
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous | Liquid, Intradermal | Total
Number analyzed (Participants) | 165 | 167 | 191 | 523
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 165 | 167 | 191 | 523
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.0 (4.4) | 26.8 (4.5) | 27.7 (4.9) | 27.2 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 80 | 102 | 263
  Male | 84 | 87 | 89 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 17 | 12 | 35
  Not Hispanic or Latino | 159 | 150 | 179 | 488
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 6 | 5 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 18 | 13 | 19 | 50
  White | 129 | 144 | 156 | 429
  More than one race | 8 | 3 | 8 | 19
  Unknown or Not Reported | 0 | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 165 | 167 | 191 | 523

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) Based on Vaccinia-specific Individual Peak Plaque Reduction Neutralization Titers (PRNT) Following 2 Doses of IMVAMUNE® Lyophilized Versus Following 2 Doses of IMVAMUNE® Liquid Administered Subcutaneously, ITT Population
Description: Blood was collected from participants for testing in the PRNT assay with vaccinia-Western Reserve (replicating vaccinia) as the assay antigen. The geometric mean titers were calculated for each participant's individual peak titer after second vaccination. Titer values below limit of detection were replaced by 7.5 (half the lower limit of detection) for analysis.
Time Frame: Days 14, 28 and 180 after 2nd vaccination
Population: The ITT analysis population for the immunogenicity summaries include all participants with results for the visit. Participants were analyzed as randomized. Not receiving the second vaccination or second vaccination being out of window was not considered.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous
Number analyzed (Participants) | 161 | 164
titer | 77.9 [62.9 to 96.5] | 46.7 [37.9 to 57.4]
Statistical Analysis 1: Comparison: Lyophilized, Subcutaneous vs Liquid, Subcutaneous; The sample size calculations targeted at least 80% power to test non-inferiority for the primary and secondary immunogenicity end points for two investigational arms in reference to a control arm. Assuming a standard deviation of 2.8 for log2 peak PRNT or ELISA titer in each group, a non-inferiority margin of 2.0-fold, a type I error rate of 1.25% (Bonferroni adjusted for 2 comparisons), and drop-out rate of 10%, 165 participants in each group were to be enrolled to achieve 148 evaluable; Test type: Non-Inferiority — The mean difference in log2 transformed peak titers between IMVAMUNE® (1x10^8 TCID50) liquid formulation (Liquid SC Group) and IMVAMUNE® (1x10^8 TCID50) lyophilized formulation (Lyophilized SC) with its associated two-sided 97.5% confidence interval (CI) was computed. If the upper limit of the 97.5% CI was less than 1, then the Lyophilized SC was considered non-inferior to the Liquid SC group. The difference and the CI are reported on the log2 scale; Mean Difference (Final Values) = -0.74, 97.5% CI 2-sided [-1.23 to -0.25]

2. Primary Outcome: GMT Based on Vaccinia-specific Individual Peak PRNT Following 2 Doses of IMVAMUNE® Lyophilized Versus Following 2 Doses of IMVAMUNE® Liquid Administered Subcutaneously, Per Protocol Population
Description: as for outcome 1
Time Frame: Days 14, 28 and 180 after 2nd vaccination
Population: The per protocol (PP) analysis population includes subjects who received two doses of vaccine in window and contributed both pre- and post-vaccination blood samples and had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous
Number analyzed (Participants) | 145 | 149
titer | 87.8 [71.2 to 108.3] | 49.5 [40.0 to 61.3]
Statistical Analysis 1: Comparison: Lyophilized, Subcutaneous vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.83, 97.5% CI 2-sided [-1.32 to -0.33]

3. Primary Outcome: GMT Based on Vaccinia-specific Individual Peak PRNT, Following 2 (Lower) Doses Liquid IMVAMUNE® Administered Intradermally Versus 2 (Higher) Doses of Liquid IMVAMUNE® Administered Subcutaneously, ITT Population
Description: as for outcome 1
Time Frame: Days 14, 28 and 180 after 2nd vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid, Intradermal | Liquid, Subcutaneous
Number analyzed (Participants) | 187 | 164
titer | 45.2 [37.0 to 55.4] | 46.7 [37.9 to 57.4]
Statistical Analysis 1: Comparison: Liquid, Intradermal vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The mean difference in log2 transformed peak titers between IMVAMUNE® (1x10^8 TCID50) liquid formulation subcutaneously (Liquid SC Group) and IMVAMUNE® (2x10^7 TCID50) formulation intradermally (Liquid ID) with its associated two-sided 97.5% confidence interval (CI) was computed. If the upper limit of the 97.5% CI was less than 1, then the Liquid ID was considered non-inferior to the Liquid SC group. The difference and the CI are reported on the log2 scale; Mean Difference (Final Values) = 0.05, 97.5% CI 2-sided [-0.43 to 0.52]

4. Primary Outcome: GMT Based on Vaccinia-specific Individual Peak PRNT, Following 2 (Lower) Doses Liquid IMVAMUNE® Administered Intradermally Versus 2 (Higher) Doses of Liquid IMVAMUNE® Administered Subcutaneously, Per Protocol Population
Description: Blood was collected from participants for testing in the PRNT assay with vaccinia-Western Reserve (replicating vaccinia) as the assay antigen. The geometric mean titers were calculated for each timepoint as well as for the peak titer after second vaccination. Titer values below limit of detection were replaced by 7.5 (half the lower limit of detection) for analysis.
Time Frame: Days 14, 28 and 180 after 2nd vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid, Intradermal | Liquid, Subcutaneous
Number analyzed (Participants) | 146 | 149
titer | 59.6 [48.1 to 74.0] | 49.5 [40.0 to 61.3]
Statistical Analysis 1: Comparison: Liquid, Intradermal vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.27, 97.5% CI 2-sided [-0.77 to 0.23]

5. Primary Outcome: Number of Participants Reporting Serious Adverse Events Associated With IMVAMUNE® Vaccination
Description: An SAE is defined as an AE or suspected adverse reaction is considered serious if, in the view of either the investigator or the sponsor, it results in death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or a congenital anomaly/birth defect. Those SAEs considered associated are those with a known temporal relationship, or the event is known to occur in association with study product or with a product in a similar class of study products AND no alternate etiology is identified.
Time Frame: Day 0 through 180 days after second vaccination
Population: The safety population includes all participants receiving at least one vaccination.
Measure: Number; unit: participants
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous | Liquid, Intradermal
Number analyzed (Participants) | 165 | 167 | 191
participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Assessed With Grade 3 and 4 Laboratory Toxicities Associated With IMVAMUNE®.
Description: Safety laboratory parameters included hemoglobin, white blood cells (WBC), platelets, ALT, and serum creatinine. These parameters were evaluated at Day 0 and 14 days after vaccination. Thresholds for Grade 3 or 4 were hemoglobin less than 8.0 g/dL, WBC less than 2000 cells/mm^3, platelets less than 50,000 cells/mm^3, ALT 5.0 times the upper limit of normal (ULN) or greater, and serum creatinine of 1.9 times ULN or greater. Associated with IMVAMUNE was defined as a known temporal relationship, or the event is known to occur in association with study product or with a product in a similar class of study products AND no alternate etiology is identified.
Time Frame: Days 0, 14 and 42
Population: The safety population includes all participants receiving at least one vaccination.
Measure: Number; unit: participants
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous | Liquid, Intradermal
Number analyzed (Participants) | 165 | 167 | 191
participants | 0 | 0 | 0

7. Secondary Outcome: GMT Based on Vaccinia-specific Individual Peak ELISA Titers, Following 2 Doses (Lower) Liquid Formulation IMVAMUNE® Administered Intradermally Versus That Obtained Following 2 Doses IMVAMUNE® Liquid Formulation Administered Subcutaneously, ITT Population
Description: Blood was collected from participants for testing in the ELISA assay with IMVAMUNE (non-replicating vaccinia in humans) as the assay antigen. The geometric mean titers were calculated for each participant's individual peak titer after second vaccination. Titer values below limit of detection were replaced by 25 (half the lower limit of detection) for analysis.
Time Frame: Days 14, 28 and 180 after 2nd vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid, Intradermal | Liquid, Subcutaneous
Number analyzed (Participants) | 187 | 164
titer | 554.0 [474.2 to 647.1] | 700.5 [595.4 to 824.1]
Statistical Analysis 1: Comparison: Liquid, Intradermal vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.34, 97.5% CI 2-sided [-0.3 to 0.71]

8. Secondary Outcome: GMT Based on Vaccinia-specific Individual Peak ELISA Titers, Following 2 Doses (Lower) Liquid Formulation IMVAMUNE® Administered Intradermally Versus That Obtained Following 2 Doses IMVAMUNE® Liquid Formulation Subcutaneously, Per Protocol Population
Description: as for outcome 7
Time Frame: Days 14, 28 and 180 after second vaccination
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Liquid, Intradermal | Liquid, Subcutaneous
Number analyzed (Participants) | 146 | 149
titer | 757.9 [664.4 to 864.6] | 769.3 [661.8 to 894.2]
Statistical Analysis 1: Comparison: Liquid, Intradermal vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Mean Difference (Final Values) = 0.02, 97.5% CI 2-sided [-0.31 to 0.35]

9. Secondary Outcome: GMT Based on Vaccinia-specific Individual Peak ELISA Titers Following 2 Doses of IMVAMUNE® Lyophilized Formulation Versus That Obtained Following 2 Doses of IMVAMUNE® Liquid Formulation Subcutaneously, ITT Population.
Description: Blood was collected from participants for testing in the ELISA assay with IMVAMUNE (non-replicating vaccinia in humans) as the assay antigen. The geometric mean titers were calculated using the individual peak titer after second vaccination. Titer values below limit of detection were replaced by 25 (half the lower limit of detection) for analysis.
Time Frame: Days 14, 28 and 180 after 2nd vaccination.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous
Number analyzed (Participants) | 159 | 164
titer | 893.5 [750.7 to 1063.5] | 700.5 [595.4 to 824.1]
Statistical Analysis 1: Comparison: Lyophilized, Subcutaneous vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.35, 97.5% CI 2-sided [-0.74 to 0.04]

10. Secondary Outcome: GMT Based on Vaccinia-specific Individual Peak ELISA Titers Following 2 Doses of IMVAMUNE® Lyophilized Formulation Versus That Obtained Following 2 Doses of IMVAMUNE® Liquid Formulation Subcutaneously, Per Protocol Population.
Description: as for outcome 9
Time Frame: Days 14, 28 and 180 after 2nd vaccination.
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous
Number analyzed (Participants) | 145 | 149
titer | 1062.4 [920.8 to 1225.8] | 769.3 [661.8 to 894.2]
Statistical Analysis 1: Comparison: Lyophilized, Subcutaneous vs Liquid, Subcutaneous; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The mean difference in log2 transformed peak titers between IMVAMUNE® (1x108 TCID50) liquid formulation (Liquid SC Group) and IMVAMUNE® (1x108 TCID50) lyophilized formulation (Lyophilized SC) with its associated two-sided 97.5% confidence interval (CI) was computed. If the upper limit of the 97.5% CI was less than 1, then the Lyophilized SC was considered non-inferior to the Lyophilized SC group. The difference and the CI are reported on the log2 scale; Mean Difference (Final Values) = -0.47, 97.5% CI 2-sided [-0.81 to -0.12]

ADVERSE EVENTS:
Time Frame: Solicited reactogenicity symptoms were collected on memory aid for 15 days after each vaccination. Non-serious unsolicited adverse events were collected for 28 days after each vaccination. Serious adverse events were collected through 180 days after the second vaccination.
Description: Reactogenicity symptoms solicited on the memory aid are counted as an event if occurring at any time during the 15 day period
Arm/Group | Lyophilized, Subcutaneous | Liquid, Subcutaneous | Liquid, Intradermal
All-Cause Mortality (participants affected / at risk) | 0/165 | 0/167 | 0/191
Serious Adverse Events (participants affected / at risk) | 1/165 | 2/167 | 1/191
Other Adverse Events (participants affected / at risk) | 164/165 | 161/167 | 191/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyophilized, Subcutaneous (N=165) | Liquid, Subcutaneous (N=167) | Liquid, Intradermal (N=191)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lyophilized, Subcutaneous (N=165) | Liquid, Subcutaneous (N=167) | Liquid, Intradermal (N=191)
Myalgia (General disorders) | 81 (108) | 69 (83) | 58 (75)
Chills (General disorders) | 31 (36) | 21 (22) | 28 (32)
Headache (Nervous system disorders) | 83 (116) | 72 (89) | 79 (110)
Nausea (Gastrointestinal disorders) | 40 (49) | 36 (42) | 44 (50)
Malaise (General disorders) | 90 (135) | 83 (112) | 98 (127)
Appetite disorder (Metabolism and nutrition disorders) | 39 (47) | 25 (28) | 39 (46) — Solicited as "Change in appetite"
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 (32) | 15 (17) | 34 (40)
Injection site pain (General disorders) | 155 (265) | 152 (265) | 125 (181)
Injection site pruritus (General disorders) | 82 (114) | 81 (110) | 170 (259)
Axillary pain (General disorders) | 25 (30) | 30 (34) | 40 (47) — Solicited as "Underarm pain"
Oedema peripheral (General disorders) | 12 (12) | 10 (11) | 20 (25) — Solicited as "Underarm swelling"
Injection site erythema (General disorders) | 128 (212) | 136 (222) | 190 (342)
Injection site swelling (General disorders) | 108 (172) | 116 (182) | 190 (337)
Vaccination Site Discolouration (General disorders) | 16 (17) | 7 (7) | 122 (183)
Vaccination Site Haematoma (General disorders) | 9 (10) | 6 (8) | 12 (16)
Vaccination Site Nodule (General disorders) | 41 (46) | 34 (41) | 35 (49)
Upper Respiratory Tract Infection (Infections and infestations) | 20 (22) | 9 (9) | 14 (14)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 4 (5) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less